CLINICAL TRIAL: NCT02429934
Title: Efficacy of Abatacept in Inflammatory Polyarthritis of Systemic Lupus Erythematosus (SLE)
Brief Title: Abatacept for SLE Arthritis (IM101-330)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Response rate in placebo group for primary outcome was 100% on interim analysis.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-330 SLE Arthritis
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Systemic Lupus Erythematosus Arthritis
Keywords: Systemic Lupus Erythematosus (SLE); Abatacept (Orencia); Arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abatacept also known as Orencia also known as CTLA4Ig (Active Comparator): 32 SLE patients to be treated with subcutaneous abatacept 125mg sq once a week for 16 weeks.
  Interventions: Biological: abatacept also known as Orencia also known as CTLA4-Ig
- Placebo (Placebo Comparator): 32 SLE patients to be treated with subcutaneous placebo once a week for 16 weeks. Injection will be vehicle injected subcutaneously once a week for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: abatacept also known as Orencia also known as CTLA4-Ig — 125mg injected subcutaneously weekly for 16 weeks
  Other Names: Orencia
  Arms: Abatacept also known as Orencia also known as CTLA4Ig
Drug: Placebo
  Arms: Placebo

SUMMARY:
This research trial is for patients who have been diagnosed with systemic lupus erythematosus (SLE) with swollen, tender joints (which is called inflammatory polyarthritis) because of the SLE.

The purpose of this clinical research study is to evaluate the safety and effectiveness of treatment with abatacept (Abatacept) 125mg injected subcutaneously (under the skin) weekly for 16 weeks versus placebo injections(a substance with no active ingredients and therefore may have no treatment benefit) in subjects with SLE and inflammatory polyarthritis. The effectiveness will be assessed primarily by the number of swollen, tender joints (called a joint count) at each of study visits.

Study Medication Abatacept is approved in the U.S. for treating rheumatoid arthritis by prescription and has not been approved by the U.S. Food and Drug Administration for treating SLE yet.

In this study, subjects will receive treatment with either abatacept or placebo once a week for 16 weeks (a total of 16 injections).

ELIGIBILITY:
Inclusion Criteria:

1. Meet at least 4 of the 11 American College of Rheumatology (ACR) 1997 criteria for classification of SLE (see Appendix 1).OR meet the recent classification recommended by SLICC (Appendix 2) 6
2. ≥3 swollen and tender joints on 2 examinations at least 2 weeks apart and no more than 8 weeks apart.
3. SLEDAI2K score ≥4 indicating active disease.
4. Documented positive ANA (≥1:80) and/or anti-dsDNA during course of SLE.
5. Men and women, at least 18 years of age. Women of childbearing potential must use adequate method(s) of contraception to avoid pregnancy throughout the study and for up to 2 months after last study drug dose. They must have a negative serum or urine pregnancy test prior to the start of study medication.
6. Background therapies allowed: antimalarials (dose constant for ≥ one month before study entry and during 16 weeks of trial), methotrexate (same criteria as for antimalarials), azathioprine (same criteria), mycophenolate (same criteria), leflunomide (same criteria).

During the screening period and for up to 6 weeks after randomization, a daily prednisone (or equivalent) regimen of up to 20 mg daily may be initiated to treat the moderate to severe disease activity present at screening. The initial steroid regimen is not required if investigators or patients believe that the risks would outweigh the potential benefits. Patients who do not take any glucocorticoids during the study will be included in the treatment groups and analysis.

*Steroids should be tapered to a target dose of no more than 10 mg/day of prednisone (or equivalent) by the end of Week 8 (Day 56). The steroid regimen should be tapered as quickly as safely possible. Prednisone dose requirements higher than 10 mg daily at the 8 week visit will cause the patient to be ruled a non-responder for the abatacept treatment arm.

Exclusion Criteria:

1. Subjects with active infection requiring oral or IV antibiotics within one month of first dose of study medication.
2. Subjects with BILAG A in any system outside the musculoskeletal system.
3. Subjects with positive quantiferon Gold test in the absence of treatment for tuberculosis.
4. Subjects with positive tests for active infection with hepatitis B or C during the past 6 months. Any confirmed positive test for HIV at any time prior to entry into this study.
5. Subjects with active glomerulonephritis (>3 g protein/24h and/or active urine sediment).
6. Subjects with active CNS disease.
7. Subjects with any other serious disease that would require immunosuppressive or parenteral anti-microbial therapy outside the study protocol.
8. Inability to self-administer subcutaneous injections, to comply with instructions, or to keep appointments for study visits.
9. Treatment with rituximab within the past 6 months (B cells must be detectable in peripheral blood at onset of treatment with study biologic), belimumab within the past 5 months, cyclophosphamide within the past 3 months.
10. Treatment with any other immunomodulatory biologic or cyclophosphamide during treatment with abatacept is not allowed.
11. Patients requiring >20 mg of prednisone daily.
12. Women who are pregnant or breast feeding.
13. Women of child bearing potential unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 2 months after last study drug.
14. Subjects with a history of cancer within the last five years (other than non-melanoma skin cell cancers cured by local resection).
15. Any laboratory test results that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10; Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bevra Hahn, M.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California
  - University of California, San Diego, San Diego, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept: abatacept: 125mg injected subcutaneously weekly for 16 weeks
- Placebo: Placebo subcutaneous injection weekly for 16 weeks
Period: Overall Study
Arm/Group | Abatacept | Placebo
Started | 15 | 13
Completed | 11 | 10
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9.0) | 40.8 (15.3) | 42.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28
education [Count of Participants; unit: Participants]
  high school | 1 | 1 | 2
  2 year college | 2 | 6 | 8
  4 year college | 4 | 1 | 5
  trade school | 1 | 0 | 1
  master's degree | 2 | 4 | 6
  professional | 2 | 1 | 3
  other | 3 | 0 | 3
insurance [Count of Participants; unit: Participants]
  PPO | 6 | 7 | 13
  HMO | 5 | 3 | 8
  Medicare | 0 | 1 | 1
  Medicaid | 3 | 2 | 5
  unknown | 1 | 0 | 1
smoking history [Count of Participants; unit: Participants]
  never smoked | 12 | 9 | 21
  past smoker | 1 | 3 | 4
  current smoker | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least a 20% Improvement From Baseline in Tender and Swollen 28 Joint Count
Description: Assessed by physical exam. Total number of joints that are both swollen and tender were assessed in each participant by a physician at each study visit.
Time Frame: Baseline, 8 Weeks, 16 Weeks
Population: subjects that completed the 8 and 16 week study visits
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 13 | 11
Participants
  8 Weeks | 11 | 11
  16 Weeks: number analyzed (Participants) | 11 | 10
  16 Weeks | 10 | 10

2. Secondary Outcome: Change in SLEDAI 2K
Description: Systemic Lupus Erythematosus Disease Activity Index (Modified in the year 2000) - The SLEDAI-2K is a modified version of a composite score based on the presence or absence of clinical signs, clinical symptoms, and immunologic laboratory results taken within 10 days of the evaluations. Each of the descriptors has a weighted score and the total score of SLEDAI-2K is the sum of all 24 descriptor scores. The total SLEDAI-2K score falls between 0 and 105, with higher scores representing higher disease activity. Decrease of 3 points in SLEDAI 2K is considered to be a clinically significant improvement.
Time Frame: Baseline, 16 weeks
Population: completers at 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Placebo subcutaneous injections weekly for 16 weeks
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale | -1.4545 (3.2669) | -3.4000 (2.8363)

3. Secondary Outcome: Change in the PGA Score
Description: Physician's Global Assessment (PGA) is a physician rating of patient's disease activity, with a range 0-3. A change of 0.8 points on a 3 point scale or less is considered as stable. Lower score means better outcome
Time Frame: Baseline, 16 weeks
Population: SLE subjects completing 16 weeks of treatment or placebo and attending the 16-week physician assessment visit.
Measure: Mean (Standard Deviation); unit: points on scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 10 | 10
points on scale | -1.3650 (3.7029) | -0.3350 (2.2289)

4. Secondary Outcome: Clinical Disease Activity Index (CDAI) Index Score
Description: CDAI is a simplified index for assessing disease activity comprising swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment), PtGA and PGA (assessed on 0-10 cm visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0-76. CDAI less than equal to (<=) 2.8 indicates disease remission, greater than (>) 2.8 to 10 = low disease activity, greater than (>) 10 to 22 = moderate disease activity, and >22 = high disease activity.
Time Frame: 16 weeks
Population: sle subjects that completed 16 week assessment visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 14.7850 (12.0459) | 14.5700 (7.9701)

5. Secondary Outcome: Synovitis, Tenosynovitis and Erosions Scores (GSUS and PDUS)
Description: Using ultrasound analysis, (Gray scale ultrasound) represents synovitis/tenosynovitis and identifies erosions. PDUS (power Doppler ultrasound) measures intensity of soft tissue inflammation by blood flow. 30 joints were evaluated using a 0 to 3 point scale for each joint and the sum of these represents PDUS. The Power Doppler Synovitis Score (PDUS) ranges from 0 to 90. Scores of 0 indicate the least amount of inflammation. A higher value of the total score for PDUS represents more severe disease level. 30 joints were evaluated using a 0 to 3 point scale for each joint and the sum of these represents GSUS. The grey scale synovial hypertrophy score (GSUS) ranges from 0 to 90. Scores of 0 indicate the least amount of inflammation of the joint. A higher value of the total score for GSUS represents more severe disease level.
Time Frame: Baseline, 16 weeks
Population: completers of 16 weeks of treatment/placebo at one study center (UCLA)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 4 | 4
score on scale
  baseline GSUS | 17.50 (7.05) | 16.00 (4.83)
  16 week GSUS | 12.75 (2.22) | 17.75 (5.19)
  baseline PDUS | 5.25 (5.12) | 1.50 (1.00)
  16 week PDUS | 2.00 (1.83) | 2.25 (1.89)

6. Secondary Outcome: Number of AEs and SAEs
Description: Total number of AEs and total number of SAEs as well as those AEs/SAEs which may be related to the study drug
Time Frame: 16 weeks
Population: All subjects dosed with either abatacept or placebo at least once.
Measure: Number; unit: adverse events
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 15 | 13
adverse events
  AEs grade II or less | 20 | 27
  AEs not related | 14 | 14
  AEs possibly related | 5 | 10
  AEs probably related | 1 | 3
  AEs grade III or higher | 1 | 0
  SAEs | 1 | 0

7. Secondary Outcome: Number of Tender and Swollen Joints
Description: Total number of joints that are both swollen and tender were assessed in each participant by a physician at each study visit
Time Frame: baseline, 4, 8, 12 and 16 weeks
Population: Each timepoint reports the number of participants who attended each visit for physician assessment
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 15 | 13
joints
  baseline | 6.73 (4.53) | 5.00 (1.41)
  week 4 | 2.80 (2.65) | 1.54 (1.10)
  week 8: number analyzed (Participants) | 13 | 11
  week 8 | 1.77 (2.13) | 0.45 (0.69)
  week 12: number analyzed (Participants) | 12 | 11
  week 12 | 1.58 (2.19) | 1.00 (1.34)
  week 16: number analyzed (Participants) | 11 | 10
  week 16 | 1.82 (2.27) | 0.50 (0.97)

8. Secondary Outcome: Change in the Total Sum of Tender and Swollen Joints
Description: as for outcome 7
Time Frame: Baseline, 16 weeks
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 11 | 10
Joints | -5.1818 (4.2619) | -4.2000 (1.3116)

9. Secondary Outcome: Number of Patients Who Tapered Prednisone to <10mg/Day
Description: This analysis is for the subset of patients who start the study taking 10 to 20mg of prednisone per day.
Time Frame: 16 weeks
Population: This analysis is for the subset of patients who start the study taking 10 to 20mg of prednisone per day. Among all the subjects entered, 6 in each group were taking 10 mg of prednisone daily or higher at baseline
Measure: Number; unit: participants
Groups:
- Placebo: placebo injected subcutaneously weekly for 16 weeks
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 6 | 6
participants | 2 | 0

10. Secondary Outcome: Mean Prednisone Dose (mg/Day)
Description: prednisone dose (mg/day) is recorded at baseline, 8 and 16 weeks for each subject being assessed at that study visit. Then a mean for all the subjects in each group at each time point was calculated.
Time Frame: Baseline, 8 and 16 weeks
Population: Results are reported for the number of participants who completed the study visit/assessment at each time point
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 15 | 13
mg per day
  baseline | 4.73 (7.73) | 4.77 (6.64)
  8 weeks: number analyzed (Participants) | 13 | 11
  8 weeks | 5.46 (7.98) | 5.64 (6.89)
  16 weeks: number analyzed (Participants) | 11 | 10
  16 weeks | 8.45 (10.04) | 5.70 (7.99)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 20 weeks after initial dose (visit 1)
Description: We used clinicaltrials.gov definitions
Arm/Group | Abatacept | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/13
Other Adverse Events (participants affected / at risk) | 6/15 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=15) | Placebo (N=13)
flare of lupus nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient developed increased proteinuria, was removed from clinical trial and treated with increased immunosuppression and problem resolved, Judged not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=15) | Placebo (N=13)
skin reaction at injection site (Skin and subcutaneous tissue disorders) | 6 (9) | 3 (4) — soreness and tenderness around point of subcutaneous injection for 1-2 days post injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02429934/Prot_SAP_000.pdf